CLINICAL TRIAL: NCT00459524
Title: Longitudinal Assessment of Neurocognitive Function and Quality of Life of Patients With Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome (MDS) Undergoing Treatment
Brief Title: Quality of Life of Patients With Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0060
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Leukemia; Quality of Life; Questionnaire; Survey; Neurocognitive Function; AML; MDS; QOL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire: AML and MDS Patients
  Interventions: Behavioral: Questionnaire; Behavioral: Neurocognitive Testing

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires taking about 30 minutes to complete.
  Other Names: Survey
Behavioral: Neurocognitive Testing — Neurocognitive testing lasting 30 minutes. Patients will be asked to complete certain tasks that require the use of their hands, eyes, and ears.

SUMMARY:
Primary Objectives:

* To compare the neuropsychiatric (NP) and neurocognitive (NC) symptoms and assess the quality of life (QOL) in older patients (age > 18) with acute myelogenous leukemia (AML) or high-risk myelodysplastic syndrome (MDS) receiving different therapies, chemotherapy (Clofarabine + ara-C) or targeted therapies (PKC412 + low-dose ara-C, or R115777 + low-dose ara-C, or decitabine, or STI + low-dose ara-C).
* To determine whether there is a correlation between the number of packed red blood cell (PRBC) transfusions and cognitive scores and/or QOL.

DETAILED DESCRIPTION:
You will participate in a series of neurocognitive tests. For these tests, you will be asked to complete certain tasks that require the use of your hands, eyes, and ears. The neurocognitive testing will take about 30 minutes.

You will answer some questionnaires about disease symptoms and your quality of life. It will take about 30 minutes to complete the questionnaires.

You will participate in these neurocognitive tests and fill out the questionnaires before you begin cancer therapy. Your interval testing will coincide with your clinic visit evaluations, which will be approximately at 1 month, 3 months, and 6 months. If you do not receive therapy, you will be asked to complete the neurocognitive tests at baseline and then again on your follow up clinic visit evaluations, which will be approximately at 3 months and at 6 months. You may be asked to continue your participation in these neurocognitive tests and fill out questionnaires approximately every 3 months thereafter.

This is an investigational study. About 306 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed AML or MDS. Patients who fail an MDS/AML therapy and receive other therapies may be asked to continue participation in this neurocognitive study.
2. Patients who are 18 years of age or older.
3. Patients who are seen in the MDACC adult Leukemia clinic. Patients who do not enroll onto therapy protocols are also eligible.
4. Patients must sign the informed consent.

Exclusion Criteria:

1) Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute myelogenous leukemia or myelodysplastic syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2004-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Effect of cancer therapy on AML or MDS patients (longitudinal assessment neuropsychiatric (NP), neurocognitive (NC) symptoms, quality of life (QOL)) | Interval testing will be approximately at 1 month, 3 months, and 6 months.

SECONDARY OUTCOMES:
Effects of therapy on the ability to think, quality of life, the ability to perform everyday tasks, and how often side effects occur. | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Christina A. Meyers, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org